CLINICAL TRIAL: NCT06844045
Title: Clinical and Implementation Outcomes of a Point of Care Sexually Transmitted Infection Testing Strategy to Improve HIV Prevention Service Delivery in Adolescents
Brief Title: Point of Care STI Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Sarah Wood, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 24-1934
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Point of Care STI Testing
Keywords: HIV Prevention; HIV Testing; HIV Pre-Exposure Prophylaxis; Gonorrhea; Chlamydia; Sexually Transmitted Infections
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Point-of-Care Tested (Experimental): Participants in the intervention arm have received point-of-care testing for sexually transmitted infections.
  Interventions: Behavioral: Gonorrhea/chlamydia Point-of-Care Testing
- Lab Tested (No Intervention): Participants in the control arm have received lab-based testing for sexually transmitted infections.

INTERVENTIONS:
Behavioral: Gonorrhea/chlamydia Point-of-Care Testing — Point-of-care testing for sexually transmitted infections.
  Arms: Point-of-Care Tested

SUMMARY:
The proposed research hypothesizes that point-of-care testing (POCT) for sexually transmitted infections (STIs) gonorrhea and chlamydia will be a feasible, acceptable, and appropriate implementation strategy for improving HIV testing and Pre-exposure prophylaxis (PrEP) delivery in youth, by increasing opportunities for clinician-patient counseling, decreasing loss to follow up, and allowing for same-day HIV prevention service provision. This hypothesis will be tested in a pragmatic non-randomized trial comparing clinical (HIV testing and PrEP counseling and prescription) and implementation (feasibility, acceptability, and appropriateness) outcomes between adolescents receiving POCT compared to laboratory-based testing at three clinics within a large pediatric health system.

ELIGIBILITY:
Inclusion Criteria:

- Patients age 16-24 years receiving POCT or lab-based GC/CT testing

Exclusion Criteria:

- Patients with known HIV or active PrEP prescriptions.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5150 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of HIV Test Completion | Day 1 - Measured on date of STI testing
  Rates of HIV test completion on the day of gonorrhea/chlamydia testing will be compared between those who receive point-of-care vs. lab-based STI testing.

SECONDARY OUTCOMES:
Number of participants who received PrEP counseling | Day 1 - Same day as STI testing encounter
  PrEP counseling will be measured using visit note data from the date of the STI testing encounter
Time to STI treatment | Time from STI diagnosis to treatment, up to 9 months
  Days between STI test order and delivery of antibiotics for STI treatment, measured using EHR data

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Wood, MD, MSHP, Principal Investigator — Mount Sinai Adolescent Health Center
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Specify Other Time Frame After the end of the award period. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Data will be findable for the research community through the NIHM Data Archive Collection.